CLINICAL TRIAL: NCT03061877
Title: The Effect of Anxiety and Depression on Treatment Response in Rheumatoid Arthritis
Brief Title: Anxiety Depression and Rheumatoid Arthritis
Acronym: ADAR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Kun Zou, PhD, Sichuan Provincial People's Hospital
Other Study IDs: SichuanPPH201701
Record Dates: First submitted 2017-02-20; First posted 2017-02-23 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Anxiety; Depression
MeSH Terms: conditions — Arthritis, Rheumatoid; Anxiety Disorders; Depression | interventions — Patient Health Questionnaire

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anxiety or depression
  Interventions: Other: Anxiety or depression
- Non-anxiety or depression

INTERVENTIONS:
Other: Anxiety or depression — The presence of anxiety or depression measured by the Hospital Anxiety and Depression Scale (HAD)
  Groups: Anxiety or depression

SUMMARY:
Anxiety and depression are highly prevalent in people with rheumatoid arthritis (RA).This study is to investigate the effect of anxiety and depression on treatment response in people with RA using observational longitudinal study design.

ELIGIBILITY:
Inclusion Criteria:

* People diagnosed with rheumatoid arthritis according to the American College Rheumatology (ACR) criteria 2010

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People diagnosed with rheumatoid arthritis according to American College Rheumatology (ACR) criteria 2010
Sampling Method: Non-Probability Sample
Enrollment: 134 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Clinical remission | 6 months
  Clinical remission defined by the Disease Activity Score 28 (DAS28) with a score less than 2.6

CONTACTS AND LOCATIONS:
Overall Officials: Kun Zou, PhD, Principal Investigator — Sichuan Provincial People's Hospital